CLINICAL TRIAL: NCT05826652
Title: The Effect of Unilateral Subcostal Transversus Abdominis Plane Block Applied as Single or Multiple Injections on Pain in Laparoscopic Cholecystectomy Operations
Brief Title: Subcostal TAP Block With Single or Multiple Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Medical Doctor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulMU Subcostal TAP Block
Record Dates: First submitted 2023-03-26; First posted 2023-04-24 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Subcostal Transversus Abdominis Plane Block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiple injection subcostal transversus abdominis plane block (Active Comparator): . The patients in multiple injection will be given three distinct injections: 10 mL of 0.25% bupivacaine above the transversus abdominis muscle adjacent to the linea semilunaris, 5 mL of 0.25% bupivacaine between the transversus abdominis and internal oblique muscles in the subcostal region above the midclavicular line and 5 mL of 0.25% bupivacaine between the transversus abdominis and internal oblique muscles in the subcostal region above the anterior axillary line.
  Interventions: Other: Multiple injection subcostal transversus abdominis plane block
- Single injection subcostal transversus abdominis plane block (Active Comparator): A single injection of 20 mL of 0.25% bupivacaine will be administered above the transversus abdominis muscle adjacent to the linea semilunaris to the patients in Group S.
  Interventions: Other: Single injection subcostal transversus abdominis plane block
- Without Block (Active Comparator): The patients in this group will not receive any block
  Interventions: Procedure: Without Block

INTERVENTIONS:
Other: Single injection subcostal transversus abdominis plane block — Single injection subcostal transversus abdominis plane block will be applied with %2,5 Marcaine 20 ml between tranvers and rectus abdominis muscle immediately next to the linea semilunaris.
  Arms: Single injection subcostal transversus abdominis plane block
Other: Multiple injection subcostal transversus abdominis plane block — Multiple injection subcostal transversus abdominis plane block will be applied with %2,5 Marcaine 5 ml between transverse and rectus abdominis muscle, 5 ml on the transverse muscle near the semilunaris and two more 5 ml volume lateral to this point near the subcostal margin.
  Arms: Multiple injection subcostal transversus abdominis plane block
Procedure: Without Block — The patients in this group will not receive block
  Arms: Without Block

SUMMARY:
It was aimed to control pain with right-sided subcostal transversus abdominis plane block application, which is performed by applying different techniques in laparoscopic cholecystectomy operations in this study. Considering that applying technique is important in this block, the results of this study can guide practitioners in this field.

DETAILED DESCRIPTION:
A total of 90 patients, aged 18 to 65 years, with American Society of Anesthesiologists (ASA) physical status I-III, scheduled for laparoscopic cholecystectomy, will be enrolled in this study. Exclusion criteria encompasse a history of allergy to local anesthetics, chronic analgesic use, psychiatric disorders, renal or hepatic dysfunction, coagulopathy, a body mass index (BMI) > 40 kg/m², and pregnancy. Patients in Group S receive a subcostal TAP block with a single injection, patients in Group T receive a subcostal TAP block with multiple injections, and patients in Group C will not receive any form of block.

Standard monitoring protocols will be implemented upon arrival in the operating theatre and heart rate (HR), mean arterial pressure (MAP), and peripheral oxygen saturation (SpO2) will be recorded during operation. Anesthesia will be induced using propofol (2 mg/kg) and fentanyl (1 μg/kg) and muscle relaxation is achieved with rocuronium (0.5 mg/kg). and maintained using sevoflurane in a 50:50 air/oxygen mixture at a flow rate of 1 L/min. Intraoperative analgesia will be provided through a remifentanil infusion at a rate of 0-0.2 μg/kg/min.

Prior to the initiation of surgery, the subcostal TAP block will be administered in Groups S and T under sterile conditions using ultrasound guidance. A single injection of 20 mL of 0.25% bupivacaine will be administered above the transversus abdominis muscle adjacent to the linea semilunaris to the left sides of the patients in Group S. The patients in Group T will be given three distinct injections to their left sides: 10 mL of 0.25% bupivacaine above the transversus abdominis muscle adjacent to the linea semilunaris, 5 mL of 0.25% bupivacaine between the transversus abdominis and internal oblique muscles in the subcostal region above the midclavicular line and 5 mL of 0.25% bupivacaine between the transversus abdominis and internal oblique muscles in the subcostal region above the anterior axillary line.

Laparoscopic cholecystectomy will be performed using four trocar placements on the right side of the abdomen. Postoperative analgesia was managed with a patient-controlled analgesia (PCA) device containing tramadol.

Postoperative remifentanil concumption will be estimated at the end of the operation. Assessments will be conducted at 30th minute, 1st, 3rd, 6st and 24th hours postoperatively, with parameters including pain, nausea, and total PCA consumption. Pain intensity will be measured using the Visual Analogue Scale (VAS; 0 = no pain, 10 = worst imaginable pain). Postoperative nausea and vomiting (PONV) will be evaluated using a verbal descriptive scale (VDS) (0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV) [10]. Patient satisfaction will beevaluated at discharge using a five-point Likert scale (1 = strongly unsatisfied, 5 = strongly satisfied). Complications, including infection, bleeding, and subcutaneous emphysema will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. ASA I-III
3. Patients scheduled for laparoscopic cholecystectomy operations

Exclusion Criteria:

1. Those who have previously had neurological and psychiatric disease symptoms and use drugs (TIA, syncope, dementia, depression, bipolar disorder, etc.)
2. Patients with known allergy to local anesthetics
3. Chronic opioid or corticosteroid users
4. Those with coagulopathy
5. Those with local or systemic infections
6. BMI>40 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Tramadol consumption | 10 minutes, 30 minutes, 1, 3, 6, 24 hours postoperatively
  Postoperative opiod consumption
Remifentanil consumption | up to 2 hours
  Intraoperative opiod consumption

SECONDARY OUTCOMES:
Visual analog scale | 30. minute
  Visual analog scale: 0 = no pain; 10 = the most severe pain you can imagine
Visual analog scale | 1. hour
  Visual ananlog scale: 0 = no pain; 10 = the most severe pain you can imagine
Visual analog scale | 3. hour
  Visual analog scale: 0 = no pain; 10 = the most severe pain you can imagine
Visual analog scale | 6. hour
  Visual analog scale: 0 = no pain; 10 = the most severe pain you can imagine
Visual analog scale | 24. hour
  Visual analog scale: 0 = no pain; 10 = the most severe pain you can imagine
Postoperative nausea and vomiting | 30. minute
  Verbal descriptive scale. 0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV
Postoperative nausea and vomiting | 1. hour
  Verbal descriptive scale:0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV
Postoperative nausea and vomiting | 3. hour
  Verbal descriptive scale:0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV
Postoperative nausea and vomiting | 6. hour
  Verbal descriptive scale:0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV
Postoperative nausea and vomiting | 24. hour
  Verbal descriptive scale:0: No PONV, 1: Mild PONV, 2: Moderate PONV, 3: Severe PONV
Patient satisfaction | 24. hour
  Five-point Likert scale: 1 = strongly unsatisfied, 5 = strongly satisfied

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University, Istanbul
  - Medeniyet University, Istanbul

IPD SHARING:
Plan to Share IPD: No